CLINICAL TRIAL: NCT01744444
Title: Treatment of Pendular Nystagmus With Gabapentin and Memantine in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012.737
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Pendular Nystagmus Patients With Multiple Sclerosis
MeSH Terms: interventions — Memantine; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine first (Experimental)
  Interventions: Drug: Memantine
- Gabapentin first (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Memantine — Patients will be randomly assigned to start on either memantine or gabapentin. For tolerance reasons, each treatment begins with a progressive increasing dose and stops with a progressive decreasing dose. The duration of the period of last dose (8 to 11 days) will be chosen according to the investigator's availability to organize post-tests.
  Arms: Memantine first
Drug: Gabapentin — Patients will be randomly assigned to start on either memantine or gabapentin. For tolerance reasons, each treatment begins with a progressive increasing dose and stops with a progressive decreasing dose. The duration of the period of last dose (8 to 11 days) will be chosen according to the investigator's availability to organize post-tests.
  Arms: Gabapentin first

SUMMARY:
Different treatment trials have been published in acquired nystagmus in the last decade; gabapentin and memantine have been found to be efficient in treating pendular nystagmus in Multiple Sclerosis. The effects of treatments are measured on nystagmus velocity, amplitude, frequency and on visual acuity. None of the trials measured a functional visual score or oscillopsia score.

The aim of our study is to evaluate the effect of gabapentin and memantine on the mean velocity, amplitude and frequency of pendular nystagmus, as well as on oscillopsia, visual acuity and vision-specific health-related quality of life score, in 10 patients with multiple sclerosis. The primary object is to find out the best variable to evaluate the efficiency of nystagmus treatment and the secondary, to compare the efficiency of both gabapentin and memantine in a common population of patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients may have a clinically definite, laboratory-supported diagnosis of multiple sclerosis according to the Mac Donald criteria.
* All patients may present a chronic acquired pendular nystagmus due to MS, observed over a period of 6 months.
* All patients will be informed about the design and purpose of the study, and all will give their informed, written consent to the protocol, which may have been approved by the local ethics committee.
* Age: above 18
* Able to understand the instructions
* Having a health coverage
* Able to sit down for 1 hour
* Stable dosage of previous medications (beginning 3 weeks previously and terminating at the end of the trial duration), except for steroids, gabapentin or memantine.

Exclusion Criteria:

* Ophthalmological

  * Other ophthalmological disorder that could impair corrected visual acuity (Maculopathy, Retinopathy…)
* Neurological

  * Ongoing seizure
  * Severe handicap that does not allow sitting down position for 1 hour
* Suicidal behavior or risk
* Treatment

  * Under memantine or gabapentin medication (these medications should have been stopped for at least 1 week for gabapentin and 3 weeks for memantine)
  * Under morphine, N-methyl-D-aspartate such as amantadine, ketamine or dextromethorphan
  * Steroid medication for a current relapse (beginning 3 weeks previously and terminating at the end of the trial duration)
  * Known hypersensitivity to memantine or gabapentin
* General

  * Unstable medical state
  * Patient with a galactose intolerance, a lapp lactase deficiency or glucose-galactose malabsorption
  * Moderate renal failure (creatinine clearance < 50 mL/min on bioassay dated from less than one month)
  * Recent heart infarction (<3months)
  * Unstable congestive heart insufficiency
  * Unstable arterial hypertension
  * Leucopenia (<2500/mm3)
  * Transaminase increase (>5 time normal values)
* Pregnancy (on questioning)
* Tutelage or any legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Velocity using eye movement recording | at Day17-21
Velocity using eye movement recording | at Day34-42
Velocity using eye movement recording | at Day64-79
Velocity using eye movement recording | at Day81-100

SECONDARY OUTCOMES:
Functional score on questioning | at Day17-21, Day34-42, Day64-79, Day81-100
Subjective measure of oscillopsia | at Day17-21, Day34-42, Day64-79, Day81-100
Far visual acuity | at Day17-21, Day34-42, Day64-79, Day81-100

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tilikete, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Neurologique Unité de Neuro-Ophtalmologie, Bron, France

REFERENCES:
- [Background] Nerrant E, Abouaf L, Pollet-Villard F, Vie AL, Vukusic S, Berthiller J, Colombet B, Vighetto A, Tilikete C. Gabapentin and Memantine for Treatment of Acquired Pendular Nystagmus: Effects on Visual Outcomes. J Neuroophthalmol. 2020 Jun;40(2):198-206. doi: 10.1097/WNO.0000000000000807. PMID 31169568